CLINICAL TRIAL: NCT05747391
Title: An Evaluation of Medical Study Experiences of Patients With Rosacea
Brief Title: Assessment of Rosacea Patients' Clinical Trial Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 83850357
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Taking part in medical trials usually favors a particular demographic group. But there is limited research available to explain what trial attributes affect the completion of these specific demographic groups.

This study will admit a wide range of data on the clinical trial experience of Rosacea patients to determine which factors prevail in limiting a patient's ability to join or finish a trial.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future Rosacea patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of Rosacea
* Ability to understand the study procedures, benefits and risks, and sign a written informed consent document.

Exclusion Criteria:

* Inability to perform regular electronic reporting
* Women who are pregnant, intend to become pregnant, or are lactating
* Enrolled in another research study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Rosacea who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to join in an Rosacea clinical study | 3 months
Number of Rosacea patients who remain in clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hopkinson D, Moradi Tuchayi S, Alinia H, Feldman SR. Assessment of rosacea severity: A review of evaluation methods used in clinical trials. J Am Acad Dermatol. 2015 Jul;73(1):138-143.e4. doi: 10.1016/j.jaad.2015.02.1121. Epub 2015 Mar 19. PMID 25799418
- [Background] Yang JH, Hwang EJ, Moon J, Yoon JY, Kim JW, Choi S, Cho SI, Suh DH. Clinical efficacy of herbal extracts in treatment of mild to moderate acne vulgaris: an 8-week, double-blinded, randomized, controlled trial. J Dermatolog Treat. 2021 May;32(3):297-301. doi: 10.1080/09546634.2019.1657792. Epub 2019 Oct 16. PMID 31424962
- [Background] Egeberg A, Weinstock LB, Thyssen EP, Gislason GH, Thyssen JP. Rosacea and gastrointestinal disorders: a population-based cohort study. Br J Dermatol. 2017 Jan;176(1):100-106. doi: 10.1111/bjd.14930. Epub 2016 Oct 31. PMID 27501017

DOCUMENTS (1):
  • Informed Consent Form (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT05747391/ICF_000.pdf